CLINICAL TRIAL: NCT03132402
Title: ELISA Validation of Hypersensitive Rapid Diagnostic Test Results for Detection of P. Falciparum Using Field Samples From Prevalence Surveys.
Brief Title: ELISA Validation of Hypersensitive Rapid Diagnostic Test Results for Detection of P. Falciparum
Acronym: ELISA
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1701
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2017-04

CONDITIONS: Plasmodium Falciparum
Keywords: Elisa; Plasmodium Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored blood samples from participants who participated in TMT protocol with sufficient volume
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ELISA validation — ELISA validation of hypersensitive rapid diagnostic test results for detection of P. falciparum

SUMMARY:
Elimination of P. falciparum (PF) malaria across a territory requires universal access to treatment of clinical cases for communities, and specific targeting of places or population groups where malaria transmission persists in spite of generalized access to treatment. In particular, a large prevalence of carriers of PF parasites is suspected to be one of the reasons for malaria persistence. The fact that these carriers are not developing symptoms allow them to harbour and transmit parasites over long periods of time. They are likely to contribute significantly the transmission in their community and even beyond it according to their movement patterns.

Identifying these pockets of high asymptomatic carriage is a key component of the malaria elimination strategy, as it allows targeting specific interventions, such as targeted mass-treatment, to quickly drain the asymptomatic reservoir.

Strategically to achieve this goal we need to be able to identify quickly and reliably the villages or groups of villages in which the asymptomatic reservoir is large and should be addressed by targeted mass drug administration (MDA).

There are no point of care tests currently available to detect asymptomatic carriers accurately. The available Rapid Diagnostic Tests (normal RDT) are designed to diagnose clinically relevant malaria infections. However their sensitivity for asymptomatic malaria carriers is low, since most of these individuals harbor parasitaemias below RDT detection thresholds. Currently, we are relying on high volume blood surveys, in which a small sample of the village population provides a 2mL venous blood sample that can be analysed by ultra-sensitive qPCR. This technique allows detecting very low parasitaemias. However it is a high cost test and technical requirements to use qPCR limit the number of samples that can be tested. In addition as the analysis must be done in a laboratory, the time needed for shipment and analysis results in delays of 4 to 8 weeks between survey and result. Surveying remote, poorly resourced areas adds to the challenge as the samples must be shipped from the field to the laboratory, on cold chain, within 24 to 48h from blood draw.

To ensure that asymptomatic individuals are diagnosed in a cost effect and feasible manner, it is vital that a more sensitive RDT is made available for use in the field. Depending on its performance, a sensitive RDT could be used for prevalence surveys to target MDA, or directly for interventions based on treatment of positive individuals (reactive case detection or mass screening and treatment).

A new hypersensitive RDT (hsRDT) has now been developed but before it can be utilised for elimination surveys we need to validate both its technical properties (sensitivity and specificity) and its usefulness in the field to detect PfHRP2 presence compared to a gold standard control ELISA (Enzyme Linked Immuno-Sorbent Assay) test. This will allow confirmation of false- and true- positive among samples.

ELIGIBILITY:
Inclusion Criteria:

* Samples from participants who participated in TMT protocol with sufficient volume to perform ELISA (minimum40 µL) and for which an hsRDT result is already available.
* Specimens have been stored at required temperature (-80 °C or below)

Exclusion Criteria:

• Specimen unsuitable for testing for any technical reasons

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: No new participants required for this study. Samples are aliquots from anonymized blood samples for which consent already given from participants participated in TMT protocol.
Sampling Method: Non-Probability Sample
Enrollment: 1656 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of hsRDT compared to ELISA (gold standard) for detection of PfHRP2 antigen | 3 months
Specificity of hsRDT compared to ELISA (gold standard) for detection of PfHRP2 antigen | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes